CLINICAL TRIAL: NCT02413567
Title: Evaluation of Duodenal Mucosal Resurfacing for the Treatment of Type 2 Diabetes
Brief Title: Evaluation of Duodenal Mucosal Resurfacing in Subjects With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-20000 A & B
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMR Procedure (Experimental): Subjects receive the endoscopic DMR procedure in this arm
  Interventions: Device: DMR Procedure (Fractyl)

INTERVENTIONS:
Device: DMR Procedure (Fractyl) — Endoscopic procedure

SUMMARY:
The purpose of this study is to evaluate the Fractyl Duodenal Mucosal Resurfacing (DMR) Procedure for the treatment of Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria

1. 28 -75 years of age
2. Diagnosed with Type 2 Diabetes for less than 10 years
3. HbA1c of 7.5 - 10.0% (59-86 mmol/mol)
4. Body Mass Index (BMI) ≥ 24 and ≤ 40 kg/m2
5. On a minimum of 1 stable oral anti-diabetic medications with no changes in medication in the previous 3 months prior to study entry
6. Willing to comply with study requirements and able to understand and comply with informed consent
7. Sign an informed consent form

Exclusion Criteria

1. Diagnosed with Type 1 Diabetes or with a history of ketoacidosis
2. Probable insulin production failure, defined as fasting C Peptide serum <1ng/mL (333pmol/l)
3. Current use of Insulin
4. Use of Glucagon like peptide (GLP)-1 analogues
5. Hypoglycemia unawareness or a history of severe hypoglycemia (at least 1 severe hypoglycemic event, as defined by need for third-party-assistance, in the last year)
6. Known autoimmune disease, as evidenced by a positive anti glutamic acid decarboxylase (GAD) test, including Celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
7. Previous gastrointestinal (GI) surgery that could affect the ability to treat the duodenum such as subjects who have had a Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions
8. History of chronic or acute pancreatitis
9. Known active hepatitis or active liver disease
10. Symptomatic gallstones or kidney stones, acute cholecystitis or history of duodenal inflammatory diseases including Crohn's Disease and Celiac Disease
11. History of coagulopathy, upper gastro-intestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia
12. Use of anticoagulation therapy (such as Warfarin) which cannot be discontinued for 7 days before and 14 days after the procedure
13. Use of P2Y12 inhibitors (clopidrogel, pasugrel, ticagrelor) which cannot be discontinued for 14 days before and 14 days after the procedure. Use of aspirin is allowed.
14. Unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during treatment through 4 weeks post procedure phase
15. Taking corticosteroids or drugs known to affect GI motility (e.g. Metoclopramide)
16. Receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
17. Persistent Anemia, defined as Hgb < 10 mg/dl
18. Estimated glomerular filtration rate (eGFR) or Modification of Diet in Renal Disease (MDRD) <30 ml/min/1,73m^2
19. Active systemic infection
20. Active malignancy within the last 5 years
21. Not potential candidates for surgery or general anesthesia
22. Active illicit substance abuse or alcoholism
23. Those who are pregnant, nursing or expect to become pregnant over the course of the study
24. Participating in another ongoing clinical trial
25. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
mean reduction in HbA1c (glycated hemoglobin) from baseline at 24 weeks post-procedure | 24 weeks post-procedure
Device or procedure related Serious Adverse Events (SAEs) and Unanticipated Adverse Device Effects (UADEs) | 24 weeks post-procedure

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (2):
  - Hopital Erasme, Brussels
  - UZ Leuven, Leuven
- Centro Clinico de Obesidad, Santiago, Chile
- Università Cattolica del Sacro Cuore, Policlinico A. Gemelli, Rome, Lazio, Italy
- Academic Medical Center, Amsterdam, Netherlands
- United Kingdom (2):
  - University College London Hospitals, London
  - King's College Hospital NHS Foundation Trust, London

REFERENCES:
- [Derived] Busch CBE, Meiring S, van Baar ACG, Gastaldelli A, DeFronzo R, Mingrone G, Hagen M, White K, Rajagopalan H, Nieuwdorp M, Bergman JJGHM. Insulin sensitivity and beta cell function after duodenal mucosal resurfacing: an open-label, mechanistic, pilot study. Gastrointest Endosc. 2024 Sep;100(3):473-480.e1. doi: 10.1016/j.gie.2024.01.031. Epub 2024 Jan 25. PMID 38280531
- [Derived] van Baar ACG, Deviere J, Hopkins D, Crenier L, Holleman F, Galvao Neto MP, Becerra P, Vignolo P, Rodriguez Grunert L, Mingrone G, Costamagna G, Nieuwdorp M, Guidone C, Haidry RJ, Hayee B, Magee C, Carlos Lopez-Talavera J, White K, Bhambhani V, Cozzi E, Rajagopalan H, J G H M Bergman J. Durable metabolic improvements 2 years after duodenal mucosal resurfacing (DMR) in patients with type 2 diabetes (REVITA-1 Study). Diabetes Res Clin Pract. 2022 Feb;184:109194. doi: 10.1016/j.diabres.2022.109194. Epub 2022 Jan 13. PMID 35032562
- [Derived] van Baar ACG, Holleman F, Crenier L, Haidry R, Magee C, Hopkins D, Rodriguez Grunert L, Galvao Neto M, Vignolo P, Hayee B, Mertens A, Bisschops R, Tijssen J, Nieuwdorp M, Guidone C, Costamagna G, Deviere J, Bergman JJGHM. Endoscopic duodenal mucosal resurfacing for the treatment of type 2 diabetes mellitus: one year results from the first international, open-label, prospective, multicentre study. Gut. 2020 Feb;69(2):295-303. doi: 10.1136/gutjnl-2019-318349. Epub 2019 Jul 22. PMID 31331994